CLINICAL TRIAL: NCT02562651
Title: Changes in Myocardial Biomechanics and Early Short-term Doxycycline Therapy in Patients With Acute Primary Anterior STEMI (ST Segment Elevation Myocardial Infarction)
Brief Title: Changes in Myocardial Biomechanics and Early Short-term Doxycycline Therapy in Patients With Primary Anterior STEMI
Acronym: MASTARD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Vyacheslav Ryabov, MD, PhD Research Institute for Cardiology, Russian Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1202
Record Dates: First submitted 2015-07-26; First posted 2015-09-29 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Vascular Diseases; Cardiovascular Diseases; Acute Myocardial Infarction
Keywords: STEMI, adverse LVR (left ventricular remodeling), MMPs, Doxycycline
MeSH Terms: conditions — Vascular Diseases; Cardiovascular Diseases; ST Elevation Myocardial Infarction; Ventricular Remodeling | interventions — Doxycycline; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxycycline (Experimental): 100 mg of Doxycycline bid for seven days in pts with STEMI underwent PCI (percutaneous coronary intervention) and with current medical therapy
  Interventions: Drug: Doxycycline
- Active comparator (Active Comparator): Standard care for STEMI
  Interventions: Other: Standard care for STEMI

INTERVENTIONS:
Drug: Doxycycline — Doxycycline bid for the first 7 days after primary anterior STEMI
  Other Names: Doxycycline Solutab
  Arms: Doxycycline
Other: Standard care for STEMI — Invasive and medical treatment for STEMI according to guidelines
  Other Names: Invasive and medical treatment for STEMI
  Arms: Active comparator

SUMMARY:
The purpose of the study is to investigate the changes of myocardial biomechanics and efficacy of doxycycline in patients with primary anterior STEMI.

DETAILED DESCRIPTION:
It is known that MMPs (matrix metalloproteinases) take part in myocardial remodeling, which lead to the adverse remodeling of left ventricular. Doxycycline inhibiting MMPs and it help to prevent collagen degradation and following LV (left ventricular) dilatation. Some experimental studies on rat models have suggested an anti-remodeling effect of doxycycline in myocardial infarction by means of decrease in activity of MMPs-2 and recovery of contractile function of myocardium. The clinical trial was performed at 2013 (D.Antoniucci), but it was a single study and confirmed theoretical and experimental background.

The study is randomized, opened, controlled. 45 patients with the first anterior STEMI will be enrolled. On admission all patients will receive reperfusion therapy during the first 24 h. Patients will be randomized by the open envelope method and after that some of the participants will be on doxycycline (100 mg b.i.d. for 7 days) in addition to routine medical therapy for STEMI, but other will be on routine medical therapy of STEMI. After that they will have echocardiography at 3-d, 7-th, 14-th days and 6 month after STEMI. The investigators will evaluate left ventricular function of these patients by routine and speckle-tracking echocardiography, incidence of cardiovascular end points (death, recurrent myocardial infarction, angina, heart failure, stroke) and their combinations, also the investigators will take blood samples to assess metalloproteinases (MMPs) and other biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 and ≤ 75 years at time of randomization (18 years and older)
* ST-elevation Q wave myocardial infarction
* term admission to an intensive care unit (ICU) in the first 24 hours of onset
* the reperfusion of the infarct-related coronary artery is not later than 24 hours after the initial onset of acute transmural myocardial infarction
* written the informed consent to participate in research

Exclusion Criteria:

* atrial fibrillation, a permanent form
* valvular heart disease
* severe comorbidity
* acute heart failure according to the Killip classification IV FC (functional class)
* history of chronic heart failure (NYHA III-IV)
* poor image quality for Echocardiography
* sinus bradycardia - heart rate of under 50 beats per minute, interventricular conduction delay (QRS > 0,11 s.) and atrioventricular block II-III degree

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Changes in LV end-diastolic volumes index, % | 14 days and 6 month after STEMI

SECONDARY OUTCOMES:
Incidence of cardiovascular death,% | 14 days and 6 month after STEMI
Incidence of the recurrent myocardial infarction,% | 14 days and 6 month after STEMI
Incidence of the angina,% | 14 days and 6 month after STEMI
Incidence of the heart failure,% | 14 days and 6 month after STEMI
Incidence of the stroke,% | 14 days and 6 month after STEMI
Incidence of the combined endpoint,% | 14 days and 6 month after STEMI
Incidence and severity of adverse events,% | 14 days and 6 month after STEMI
Changes in 2 D global longitudinals strain,Δ % | 14 days and 6 month after STEMI
Changes in MMPs and their inhibitors, other biomarkers, pg/ml | 14 days and 6 month after STEMI

CONTACTS AND LOCATIONS:
Overall Officials: Vyacheslav Ryabov, MD,PhD, Principal Investigator — Research Institute for Cardiology
Locations (1):
- Research Institutite for Cardiology, Tomsk, Tomskii Region, Russia